CLINICAL TRIAL: NCT03078504
Title: Hemodynamic Effects of Blood Flow Variation in Continuous Renal Replacement Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit patients further
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Zafar Jamkhana, MD, Associate Professor, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26817
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Acute Kidney Injury; End-stage Renal Disease
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental arm (Experimental): The patients will have the blood flow rate adjusted on CRRT gradually increased to assess the effect on hemodynamics
  Interventions: Device: continuous renal replacement therapy using System One (TM) setup (Nxstage)

INTERVENTIONS:
Device: continuous renal replacement therapy using System One (TM) setup (Nxstage) — Participants who have been prescribed continuous renal replacement therapy will have hemodynamic parameters measured at various blood flow rates
  Other Names: NxStage

SUMMARY:
Purpose of this study is to evaluate the short-term hemodynamic effects of changes in blood flow rates in critically ill patients receiving continuous renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* Acute renal failure or end-stage renal disease necessitating CRRT
* Admitted to the MICU service
* If on vasopressor/inotropic agent, norepinephrine as only intravenous pressor
* If on vasopressor/inotropic agent, at stable pressor dose for at least four hours
* If on IV fluids, stable dose of crystalloids <= 100cc/hour and is not receiving colloids for 4 hours or more prior to initiation of CRRT
* Mean arterial pressure (MAP) >= 65
* Arterial catheter present for continuous blood pressure monitoring
* CRRT duration of 48 hours or less using NxStage System One dialysis system
* successfully tolerated CRRT for at least 4 hours without clotting or hemodynamic instability
* no other procedures, blood products transfusion, or additional medication administration are anticipated during the study period

Exclusion Criteria:

* listed for organ transplant
* atrial fibrillation, other irregular heart rhythm, unstable arrhythmia
* need for more than one intravenous vasopressor agent
* intravenous vasopressor/inotropic agent other than norepinephrine (ie dobutamine, dopamine, vasopressin, epinephrine)
* therapeutic anticoagulation being administered
* known acute myocardial infarction as defined by elevated troponin along with a documented clinical diagnosis during current hospitalization
* known acute stroke, intracerebral hemorrhage, intracranial mass effect, or elevated intracranial pressure within the last 30 days.
* dialysis catheter malfunction and unable to maintain target blood flow rate
* fluid removal (ultrafiltration) rate > 100mL/hour

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zafar Jamkhana, MD, Principal Investigator — Associate Professor
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6
mean arterial pressure [Mean (Standard Deviation); unit: mmHg] | 79 (12)

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Change
Description: Change in mean arterial pressure from period 1 to period 2
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
mmHg | -0.2 (2)

ADVERSE EVENTS:
Time Frame: 40 minutes
Arm/Group | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT03078504/Prot_SAP_000.pdf